CLINICAL TRIAL: NCT04596748
Title: Prospective Randomized Double-Blind Placebo-Controlled Study of Oral Probiotics on the Microbiome and Lipidome in Acne Vulgaris
Brief Title: Oral Probiotics on the Microbiome and Lipidome in Acne Vulgaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Microbiome labs (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, Principal Investigator, Integrative Skin Science and Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISSR-Prob-GutSkin
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; skin; dermatology; acne; microbiome; probiotics
MeSH Terms: conditions — Acne Vulgaris | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be taking a placebo supplement that they will be taking by mouth once per day.
  Interventions: Dietary Supplement: Placebo
- Probiotic (Experimental): Participants will be taking a probiotic supplement that they will be taking by mouth once per day.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Bacillus Subtilis, Bacillus Clausii, Bacillus Coagulans, Bacillus Indicus HU36, MCC 102
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo caps
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine how probiotics affect sebum production and gut health in those with acne vulgaris.

DETAILED DESCRIPTION:
Probiotics have been shown in previous pilot studies to be helpful in acne and this study aims to examine how the gut microbiome and skin biophysical properties are shifted in those with acne vulgaris. In particular, this study will assess the influence of oral spore based probiotics on the skin sebum production and will assess how probiotics influence the gut microbiome and the blood levels of short chain fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 13-45
* Subjects with acne vulgaris as diagnosed by a board-certified dermatologist,having mild-moderate acne on the face with an IGA score of 2-3 and 10+ inflammatory lesions on face and 15+ total lesions.
* Subjects should experience new acne lesions on a recurrent basis within last 6 months
* Must be willing to comply with all protocol requirements
* Must be willing to have flash photo facial images taken with the imaging systems
* Males must be willing to shave any facial hair

Exclusion Criteria:

* Any systemic antibiotics used to treat acne (injected or oral)within 6 months of starting study. Any 14-day or shorter course of systemic antibiotics (injected or oral) used to treat conditions other than acne within 1 month of starting study
* Any topical antibiotic or benzoyl peroxide within 1 month of starting study or any subject unwilling to refrain from washout of topical antibacterial or benzoyl peroxide ingredient.
* Any oral probiotic or prebiotic supplementation within past 1 month
* Subjects must have no history of malignancy or cancer or diagnosis of gastrointestinal inflammatory diseases, no history or diagnosis of epilepsy, no history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis)
* Has a condition or is on medication the investigator and/or designee believe could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results
* Women who have been pregnant in the last three months, are pregnant, preparing to be pregnant or lactating, or post-menopausal.
* Is participating in a concurrent clinical research study or has participated in acne or other facial study at this or any other facility in the past 4 weeks
* Those with BMI higher than 35kg/m²
* Those that have undergone a change in hormonally based therapies, such as but not limited to oral contraceptive pills or progesterone based pills within the last two months. Progesterone releasing IUDs and spironolactone are considered hormone-based therapy.
* Commencement of a new diet (such as the ketogenic diet)or supplements within the 1 month prior to initiating participation, at the discretion of the investigator.
* Use of medications that alter blood lipids, such as statins and anti-hyperlipidemic medications
* Is participating in or has participated in acne or other facial study at this or any other facility in the past 4 weeks. Participation in survey-based studies are approved at the discretion of the investigator.
* Has a skin disease on face, other than acne, that will interfere with image collection and assessment in the opinion of the investigator
* Refusal to shave or remove facial hair that may interfere with image collection and assessment.
* Severe acne or nodulocystic acne, at the discretion of the investigator
* Use of isotretinoin within the 6 months prior to starting in study.
* Persons unwilling to avoid the following during the 4 weeks prior and during the duration of the study: self-tanning, spa tanning, or artificial tanning.
* Known allergy or irritation to the supplement or facial products utilized in the study
* Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco
* Prisoners
* Adults unable to consent

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Microbiota Diversity | 12 weeks
  Evaluation of alpha diversity
Short chain fatty acids | 12 weeks
  Blood plasma
Blood acetate levels | 12 weeks
  Blood plasma

SECONDARY OUTCOMES:
Gut microbiome changes | 4 weeks and 8 weeks
  Evaluation of alpha diversity
Change in skin microbiome | 12 weeks
  Relative abundance cutibacterium genera
Safety assessments for GI distress | 4 weeks, 8 weeks, 12 weeks
  Self assessment using Digestive Questionnaire
Change in sebum excretion rate | 4 weeks, 8 weeks, 12 weeks
  Sebumeter: 0-150 micrograms/cm^2
Change in skin hydration | 4,8 and 12 weeks
  Moisturemeter: 0-150
Change in skin pH | 4,8, and 12 weeks
  Use of pH meter
Facial redness - Image based | 4,8,12 weeks
  BTBP Clarity Mini 3D camera
Facial skin tone - Image based | 4,8,12 weeks
  BTBP Clarity Mini 3D camera
Subjective assessment of the skin | 4,8,12 weeks
  Self-assessment through Dermatology Quality of Life questionnaire
Safety assessment of acne | 4, 8, 12 weeks
  Evaluation of acne to assess for flares
Gut Microbiome Changes | 4, 8, 12 weeks
  Relative abundance of Akkermansia muciniphila

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No